CLINICAL TRIAL: NCT04179422
Title: Nutritional Status and Family Strategies Linked to Feeding in Children and Adolescents With Cerebral Palsy.
Brief Title: Nutritional Status and Family Strategies in Children With Cerebral Palsy.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, Eduardo Cuestas, Principal Investigator, National Council of Scientific and Technical Research, Argentina
Other Study IDs: IS002377
Record Dates: First submitted 2019-10-17; First posted 2019-11-27 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy; Nutrition Disorders; Child
MeSH Terms: conditions — Cerebral Palsy; Nutrition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: anthropometric measurement — weight, height, BMI
Other: nutritional questionnaire — 24hs food recall, presence of feeding disorders

SUMMARY:
Cerebral palsy (CP) is one of the neurological disorders that most often generates disability in pediatric age. Children with CP have a very high nutritional risk since their motor dysfunction causes coordination dysfunction in the processes of sucking, chewing and swallowing, which lead to insufficient intake. There are other difficulties in relation to feeding, such as the time required for feeding and the presence of gastrointestinal disorders. In addition, the families of children with CP develop different strategies that allow them to face reality. This research plan seeks to investigate the relationships between the nutritional status of children and adolescents with CP, food intake and family behavior according to the strategies they develop. This study will be observational, cross-sectional descriptive. The population will consist of children and adolescents from 2 to 18 years 11 months with a diagnosis of CP and their families attending health institutions in Córdoba. The minimum sample size in 187 subjects was calculated for an expected prevalence of 25% of feeding difficulties for an alpha 0.05 and a beta 0.20. It will be a successive sampling, until the desired sample is completed. The variables studied will be: age, weight, height, nutritional status, sex, type of CP, caloric and macro nutrient intake, type and feeding time, clinical difficulties related to feeding and family strategies For data analysis, normal continuous variables will be described in means with their standard deviations, with non-normal distribution in medians with their interquartile ranges. The daily food intake and macro nutrients will be calculated using the Food Analysis and Registration System software (SARA1.2.25). The relationship between the average energy intake, the nutritional status of children with CP and family strategies will be described. Interpretation of the data will be carried out, showing the relationship between the different areas, analyzing the connectivity of the ideas with the nutritional status.

DETAILED DESCRIPTION:
This research was an observational, descriptive, cross-sectional study. The population was made up of children and adolescents from 2 to 18 11 months years of age with CP diagnosis and their families who attended public and private health institutions in the City of Córdoba. A non-probability sequential sampling was carried out. The sample size was calculated for an expected prevalence of at least 25% of nutritional deficit in children and adolescents with CP to detect the strategies that predict good nutritional status with an odds ratio of at least 2 in 94 patients (Ortega Calvo and Cayuela Dominguez 2002) The families were invited to participate through the directors or managers of the educational centers or institutions. They were communicated orally and then in writing what the project was about.

This study included all children of both sexes from 2 to 18 years and 11 months with a diagnosis of CP defined as a disability that describes a group of permanent developmental disorders of movement and posture, which cause activity limitation, attributable to non-progressive alterations that occur in the developing fetal or infant brain. CP motor disorder is often accompanied by disturbances in sensation, perception, cognition, communication, and behavior; due to epilepsy and secondary musculoskeletal problems, who attend rehabilitation centers or public and private therapeutic educational centers in the city of Córdoba and neighboring towns that agree to participate and whose parents, guardians or caregivers sign the informed consent and want to participate. The CP diagnosis was taken from the Unique Certificate of Disability and in those children who were not established, the medical records were searched.

The normality of the continuous data was tested with the Kolmogorov-Smirnov test and they were reported as mean and standard deviations, while the non-normal distribution as medians with their interquartile ranges. Discrete data were expressed in absolute frequencies and percentages with 95% CI. The data that were non-parametric underwent a logarithmic transformation for their conversion to parametric.

The nutritional assessment, in accordance with the WHO reference parameters, was performed using the WHO Anthro Plus V1.0.4 anthropometric assessment program which uses the official WHO 2007 reference standards, providing accurate z-score values. Due to the fact that the growth patterns of the WHO (2007) do not present weight-for-age data up to 18 years of age, it was decided to use the Argentine references of the Argentine Society of Pediatrics, standardizing the weight by sex and age (2013).

Then a) Bivariate analysis will be carried out: The relationship between energy and macronutrient intake, factors related to food and nutritional assessment of children with CP, were analyzed using Chi-square tests with Fisher's test, t-test, or Mann-Whitney, as applicable. Variables that were significant with a p value <0.05 were placed in a multivariate model. b) Multivariate analysis: A multiple logistic regression model was used to identify significant predictors for adequate caloric and macronutrient intake, adjusted for sex, age, and CP severity.

The study of nutrition in patients with CP is an emerging field that has not yet been developed in our country, for which this work plan seeks to develop methodologies that promote social inclusion by making substantial and necessary contributions to improve the treatment and quality of life of children and adolescents with CP.

ELIGIBILITY:
Inclusion Criteria:

* Children with diagnosis of cerebral palsy

Exclusion Criteria:

* children with endocrine or metabolic disorders, genetic diseases and other congenital anomalies that affect or have affected their growth or nutritional status.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population of this study will be made up of children aged 2 to 18 years with a diagnosis of CP who attend public and private health institutions in Argentina.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | 2 years
  Weigth (Kg), height (cm), BMI (Kg/cm2)
feeding disorders | 2 years
  Questionnaire: number of participants with dysphagia, number of participants with sialorrhea, number of participants with constipation, number of participants with gastroesophageal reflux

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Cuestas, PhD MD, Study Director — Instituto de Investigaciones en Ciencias de la Salud
Locations (1):
- Instituto de Investigaciones en Ciencias de la Salud, Argentina, Córdoba, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
the research group is yet not decided to make individual participant data available, we wont to have a bigger data base to decide.

REFERENCES:
- [Background] Day SM, Strauss DJ, Vachon PJ, Rosenbloom L, Shavelle RM, Wu YW. Growth patterns in a population of children and adolescents with cerebral palsy. Dev Med Child Neurol. 2007 Mar;49(3):167-71. doi: 10.1111/j.1469-8749.2007.00167.x. PMID 17355471
- [Background] Bell KL, Davies PS. Prediction of height from knee height in children with cerebral palsy and non-disabled children. Ann Hum Biol. 2006 Jul-Aug;33(4):493-9. doi: 10.1080/03014460600814028. PMID 17060071
- [Result] Brooks J, Day S, Shavelle R, Strauss D. Low weight, morbidity, and mortality in children with cerebral palsy: new clinical growth charts. Pediatrics. 2011 Aug;128(2):e299-307. doi: 10.1542/peds.2010-2801. Epub 2011 Jul 18. PMID 21768315